CLINICAL TRIAL: NCT04188288
Title: Neurofeedback in Individuals With Substance Use Disorders
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to low enrollment from the COVID interruption.
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2000025618; 1K01DA039299-01A1 (NIH)
Record Dates: First submitted 2019-12-03; First posted 2019-12-05 (Actual); Results first posted 2024-09-25 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-09

CONDITIONS: Opioid-Related Disorders
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants will be blinded as to whether they are receiving experimental or control neurofeedback.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Neurofeedback (Experimental): Three imaging (fMRI) sessions of experimental feedback.
  Interventions: Device: Experimental feedback; Device: fMRI
- Control feedback (Other): Three imaging (fMRI) sessions of control feedback.
  Interventions: Device: Control feedback; Device: fMRI

INTERVENTIONS:
Device: Experimental feedback — Participants provided with feedback of target brain activation patterns (for example, in the form of a line graph) and will be instructed to try to make the line go up or down.
  Arms: Neurofeedback
Device: Control feedback — Participants provided with control type of feedback (for example, in the form of a line graph) and will be instructed to try to make the line go up or down.
  Arms: Control feedback
Device: fMRI — fMRI will be used to assess brain activity

SUMMARY:
The aim of this study is to train individuals with opioid use disorder to control their brain activity in a way that has been associated with their symptoms. Participants in the experimental group will be given direct feedback regarding their brain activity while they are undergoing functional magnetic resonance imaging (fMRI) scanning, and will try to learn to control their brain activity during these feedback sessions. A separate group of participants will be given a control form of feedback that we do not believe can have clinical benefits. Our primary hypothesis is that the neurofeedback training will reduce opioid use and clinical features of opioid use disorder more than the control feedback.

ELIGIBILITY:
Inclusion Criteria:

1. non-methadone opioid positive urine screen (as assessed during standard treatment) or indicated via Utox or self-reported past-month opioid use at screening
2. Diagnostic and Statistical Manual of Mental Disorders (DSM)-5 criteria for opioid use disorder, as assessed via structured clinical interview (SCID)
3. ≥3 months of methadone treatment

Exclusion Criteria:

1. Having any current neurologic or psychiatric disorders including current moderate to severe other DSM-5 substance use disorders with the exceptions of opioids, cocaine, tobacco and cannabis, as assessed using the SCID.
2. Failure to pass a magnetic resonance imaging (MRI) screening
3. Having significant underlying medical conditions requiring medications.
4. Women who are pregnant or nursing
5. Baseline scanning with excessive motion based on frame to frame displacement

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-03-15 (Actual); Study Completion 2023-03-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen Garrison, PhD, Principal Investigator — Yale University
Locations (1):
- Yale New Haven Hospital, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 12 participants enrolled with one participant excluded prior to randomization
Groups:
- Control Feedback: Three imaging (fMRI) sessions of control feedback.
  Control feedback (sham): Participants provided with control type of feedback (for example, in the form of a line graph) and will be instructed to try to make the line go up or down.
Period: Overall Study
Arm/Group | Neurofeedback | Control Feedback
Started | 8 | 3
Completed Scan Day 1 | 7 | 3
Completed Scan Day 2 | 5 | 3
Completed Scan Day 3 | 4 | 3
Completed Scan Day 4 | 4 | 3
Completed Scan Day 5 | 2 | 3
Completed 1 Month Follow up | 3 | 3
Completed | 3 | 3
Not Completed | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Neurofeedback | Control Feedback | Total
Number analyzed (Participants) | 8 | 3 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 3 | 11
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 1 | 6
  Male | 3 | 2 | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 7 | 3 | 10
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 8 | 3 | 11
Opioid Craving Scale [Mean (Standard Deviation); unit: score on a scale] — This outcome will be measured with the Opioid Craving Scale, a 3-item measure of craving that uses a 0-10 analog scale. Total possible score is 0-30, with higher score indicating more craving.
  score on a scale | 17.4 (7.6) | 16.8 (7.6) | 17.2 (7.2)
Quick Inventory of Depressive Symptomatology [Mean (Standard Deviation); unit: score on a scale] — This is a 16-item measure, using a 0-3 scale for each item. Total possible score is 0-48, with higher scores indicating greater symptom severity.
  score on a scale | 9.0 (5.4) | 8.7 (4.9) | 8.9 (5)

OUTCOME MEASURES:

1. Primary Outcome: Opioid Use: Urine Tests
Description: Opioid use will be monitored by weekly urine test. This will be assessed as the percentage of negative tests.
Time Frame: Baseline (week 1) to one month post follow-up (week 9)
Population: One participant in the experimental group did not have any urine tests.
Measure: Number; unit: percentage of negative tests
Units Other Than Participants: urine tests
Arm/Group | Neurofeedback | Control Feedback
Number analyzed (Participants) | 7 | 3
Number analyzed (urine tests) | 12 | 5
percentage of negative tests | 17.9 | 0

2. Primary Outcome: Opioid Use: Timeline Followback Method (TLFB)
Description: Opioid use assessed using the timeline followback method (TLFB). TLFB asks subjects to estimate drug use during a specific time period in the past. Number of participants positive or negative for drug use.
Time Frame: Baseline (week 1) to one month post follow-up (week 9)
Population: Results presented here are for participants that had completed TLFB at both baseline and follow up.
Measure: Count of Participants; unit: Participants
Arm/Group | Neurofeedback | Control Feedback
Number analyzed (Participants) | 2 | 2
Participants
  Baseline: Negative | 1 | 1
  Baseline: Positive | 1 | 1
  Follow up: Negative | 0 | 0
  Follow up: Positive | 2 | 2

3. Secondary Outcome: Mean Change in Functional Connectivity Patterns in the Brain
Description: This outcome will be assessed with functional magnetic resonance imaging (fMRI) scans. Opioid abstinence network connectivity strength will be calculated during resting state (H2a). (Data was not able to be collected at MIDT and Stroop tasks as intended.) 0 represents no engagement of the opioid abstinence network. As as a novel brain network measure, there are no defined clinical cutoffs for functional connectivity. Reported is the Z-score Fisher transformed correlation coefficient.
Time Frame: Baseline (week 1) through follow up (week 5)
Population: Results are reported for resting state as task data was not able to be collected as planned and for participants that completed all 5 scans.
Measure: Mean (Standard Deviation); unit: Fisher Z-transform corr. coefficient
Arm/Group | Neurofeedback | Control Feedback
Number analyzed (Participants) | 2 | 3
Fisher Z-transform corr. coefficient | -11.2 (13.4) | 38.7 (67.7)

4. Secondary Outcome: Mean Opioid Craving Score
Description: This outcome will be measured with the Opioid Craving Scale, a 3-item measure of craving that uses a 0-10 analog scale. Total possible score is 0-30, with higher score indicating more craving.
Time Frame: Baseline (week 1) to one month post follow-up (*week 9*)
Population: Results presented here is for participants that have both baseline and follow up data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neurofeedback | Control Feedback
Number analyzed (Participants) | 2 | 3
score on a scale
  Baseline | 18.8 (7.9) | 16.8 (7.6)
  Follow up | 23.8 (5.5) | 16.0 (4.9)

5. Secondary Outcome: Negative Affect Mean Score
Description: This outcome will be measured by the Quick Inventory of Depressive Symptomatology. This is a 16-item measure, using a 0-3 scale for each item. Total possible score is 0-48, with higher scores indicating greater symptom severity.
Time Frame: Baseline (week 1) to one month post follow-up (week 9)
Population: Results presented here is for participants that have both baseline and follow up data.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Neurofeedback | Control Feedback
Number analyzed (Participants) | 2 | 3
score on a scale
  Baseline | 12 (1.4) | 8.7 (4.9)
  Follow up | 14.5 (2.1) | 6.7 (2.5)

ADVERSE EVENTS:
Time Frame: 2 months
Description: No adverse events and/or serious adverse events took place.
Arm/Group | Neurofeedback | Control Feedback
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/3
Other Adverse Events (participants affected / at risk) | 0/8 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-10-11): https://cdn.clinicaltrials.gov/large-docs/88/NCT04188288/Prot_SAP_001.pdf
  • Informed Consent Form (2022-10-11): https://cdn.clinicaltrials.gov/large-docs/88/NCT04188288/ICF_000.pdf